CLINICAL TRIAL: NCT01253174
Title: Open-label, Randomized, Three-fold Crossover Study to Investigate the Bioequivalence of Two Different Tablet Formulations Containing 0.03 mg Ethinylestradiol (EE) and 3 mg Drospirenone (DRSP) Without [SH T470FA] and With [SH T04532A] 0.451 mg Metafolin®, and to Investigate the Bioequivalence of Two Different Tablet Formulations Containing 0.451 mg Metafolin® Without [SH T04532C] and With 0.03 mg EE/ 3 mg DRSP [SH T04532A] in 42 Healthy Young Women
Brief Title: Investigation of Bioequivalence of Ethinylestradiol (EE) and Drospirenone (DRSP) in Two Different Tablet Formulations: Yasmin and Yasmin + Levomefolate Calcium (Metafolin) & L-5-MTHF in Two Different Tablet Formulations: Levomefolate Calcium (Metafolin) and Yasmin + Levomefolate Calcium (Metafolin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 91457; 2005-001913-16 (EudraCT Number)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone; drospirenone and ethinyl estradiol combination; levomefolate calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) (Experimental): single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP)
  Interventions: Drug: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131)
- EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) (Experimental): single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca])
  Interventions: Drug: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
- L-5-MTHF Ca 0.451 mg (Metafolin) (Active Comparator): single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca])
  Interventions: Drug: L-5-MTHF Ca 0.451 mg (Metafolin)

INTERVENTIONS:
Drug: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) — single oral administration of 1 coated tablet SH T470FA (Yasmin, film-coated tablets with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP)
  Arms: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131)
Drug: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) — single oral administration of 1 coated tablet SH T04532A (film-coated tablet with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin
  Arms: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Drug: L-5-MTHF Ca 0.451 mg (Metafolin) — single oral administration of 1 coated tablet SH T04532C, containing 0.451 mg Metafolin
  Arms: L-5-MTHF Ca 0.451 mg (Metafolin)

SUMMARY:
The purpose of this study is to examine and compare the uptake of Yasmin (oral contraceptive containing drospirenone and ethinylestradiol) with or without levomefolate calcium (Metafolin, a registered vitamin supplement) in the body and to examine and compare the uptake of levomefolate calcium with or without Yasmin in the body, in healthy volunteers not using hormonal contraception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer
* Age: 18 - 38 years inclusive
* Body mass index (BMI)1: ≥ 19 and < 28 kg/m²
* Regular cyclic menstrual periods at screening OR when using combined oral contraceptives during the recruitment period reporting of natural cyclic menstrual periods prior to their use
* Willingness to use non-hormonal methods of contraception during the complete trial OR previous tubal ligation

Exclusion Criteria:

* incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, excretion and effect of the study drugs will not be normal
* known or suspected sex-steroid influenced malignancies
* endometrial hyperplasia; genital bleeding of unknown origin; uterus myomatosus
* known or suspected tumors of the liver and pituitary
* presence or history of severe hepatic disease as long as liver function values have not returned to normal
* severe renal insufficiency or acute renal failure
* thrombophlebitis, venous / arterial thromboembolic diseases; presence or history of prodromi of a thrombosis
* other conditions that increase susceptibility to thromboembolic diseases
* known neuropsychiatric diseases, especially known or suspected epilepsy, and/ or deficient status of folate or vitamin B12
* use of any other medication within 2 cycles before first study drug administration which could affect the study aim
* use of potassium sparing drugs; use of folic acid containing supplements or medicines or use of any medication within 2 cycles before first study drug administration known to interfere with folate metabolism
* inadequate folate and/or Vitamin B12 status , clinically relevant deviations in red cell folate concentrations

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Scope International, Hamburg, Hamburg, Germany

REFERENCES:
- [Result] Wiesinger H, Eydeler U, Richard F, Trummer D, Blode H, Rohde B, Diefenbach K. Bioequivalence evaluation of a folate-supplemented oral contraceptive containing ethinylestradiol/drospirenone/levomefolate calcium versus ethinylestradiol/drospirenone and levomefolate calcium alone. Clin Drug Investig. 2012 Oct 1;32(10):673-84. doi: 10.1007/BF03261921. PMID 22909145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy young women, aged 18 - 38 years inclusive, who were nonsmokers were enrolled from 16 August 2006 to 4 July 2007 at one center in Germany.
Pre-assignment Details: 147 female volunteers were screened according to the inclusion and exclusion criteria to determine that the volunteer was in a good state of health and appropriate for inclusion in the study, and 48 volunteers were randomized at one center.
Groups:
- Treatment Sequence A: Yasmin, EE30/DRSP/L-5-MTHF Ca, Metafolin: Yasmin for Period 1; EE30/DRSP/L-5-MTHF Ca for Period 2; Metafolin for Period 3. Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP) / EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]).
- Treatment Sequence B: Yasmin, Metafolin, EE30/DRSP/L-5-MTHF Ca: Yasmin for Period 1; Metafolin for Period 2; EE30/DRSP/L-5-MTHF Ca for Period 3. Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP) / Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]).
- Treatment Sequence C: EE30/DRSP/L-5-MTHF Ca, Yasmin, Metafolin: EE30/DRSP/L-5-MTHF Ca for Period 1; Yasmin for Period 2; Metafolin for Period 3. EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP) / Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]).
- Treatment Sequence D: EE30/DRSP/L-5-MTHF Ca, Metafolin, Yasmin: EE30/DRSP/L-5-MTHF Ca for Period 1; Metafolin for Period 2; Yasmin for Period 3. EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP).
- Treatment Sequence E: Metafolin, Yasmin, EE30/DRSP/L-5-MTHF Ca: Metafolin for Period 1; Yasmin for Period 2; EE30/DRSP/L-5-MTHF Ca for Period 3. Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP) / EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]).
- Treatment Sequence F: Metafolin, EE30/DRSP/L-5-MTHF Ca, Yasmin: Metafolin for Period 1; EE30/DRSP/L-5-MTHF Ca for Period 2; Yasmin for Period 3. Metafolin: single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / EE30/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca]) / Yasmin: single oral administration of 1 film-coated SHT470FA tablet (Yasmin with ethinylestradiol (EE) as free steroid), containing 0.030 mg EE + 3 mg drospirenone (DRSP).
Period: Period 1
Arm/Group | Treatment Sequence A: Yasmin, EE30/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: Yasmin, Metafolin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE30/DRSP/L-5-MTHF Ca, Yasmin, Metafolin | Treatment Sequence D: EE30/DRSP/L-5-MTHF Ca, Metafolin, Yasmin | Treatment Sequence E: Metafolin, Yasmin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE30/DRSP/L-5-MTHF Ca, Yasmin
Started | 6 | 10 | 9 | 7 | 9 | 7
Completed | 6 | 9 | 8 | 7 | 8 | 7
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Randomized but not treated | 0 | 1 | 1 | 0 | 1 | 0
Period: Period 2
Arm/Group | Treatment Sequence A: Yasmin, EE30/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: Yasmin, Metafolin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE30/DRSP/L-5-MTHF Ca, Yasmin, Metafolin | Treatment Sequence D: EE30/DRSP/L-5-MTHF Ca, Metafolin, Yasmin | Treatment Sequence E: Metafolin, Yasmin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE30/DRSP/L-5-MTHF Ca, Yasmin
Started | 6 | 9 | 8 | 7 | 8 | 7
Completed | 6 | 9 | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence A: Yasmin, EE30/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: Yasmin, Metafolin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE30/DRSP/L-5-MTHF Ca, Yasmin, Metafolin | Treatment Sequence D: EE30/DRSP/L-5-MTHF Ca, Metafolin, Yasmin | Treatment Sequence E: Metafolin, Yasmin, EE30/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE30/DRSP/L-5-MTHF Ca, Yasmin
Started | 6 | 9 | 7 | 7 | 8 | 7
Completed | 6 | 8 | 6 | 7 | 7 | 7
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants treated
Arm/Group | Entire Study Population
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Concentration (Cmax) of EE Incl. Bioequivalence (BE) Evaluation
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: up to 96 hours after administration
Population: Note that not all samples were evaluable for each outcome measure. Therefore the number of participants analyzed not necessarily matches the number of completers.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca): single oral administration of 1 film-coated SHT04532A tablet (with ethinylestradiol (EE) as clathtrate), containing 0.030 mg EE + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca])
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 42 | 42
pg/mL | 58.5 [53.1 to 64.4] | 61.6 [56.6 to 67.0]
Statistical Analysis 1: Comparison: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) vs EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca); 41 volunteers qualified for statistical analysis of BE whereas all 42 volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — A sample size of 6 volunteers per sequence was considered sufficient to establish bioequivalence, id est the 90%-confidence interval for the mean ratio is located completely within the equivalence interval limits of 80% and 125%; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 102.26, 90% CI [96.65 to 108.20] — Point estimate for the ratio [(EE30/DRSP/L-5-MTHF Ca) / Yasmin]. Bioequivalence is established if the 90% confidence interval fall within the equivalence interval limits of 80-125%

2. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of EE Incl. Bioequivalence (BE) Evaluation
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample
Time Frame: up to 96 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg∙h/mL
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 42 | 42
pg∙h/mL | 573 [521 to 632] | 595 [544 to 651]
Statistical Analysis 1: Comparison: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) vs EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 101.13, 90% CI [97.65 to 104.75] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Maximum Concentration (Cmax) of DRSP Incl. Bioequivalence (BE) Evaluation
Description: as for outcome 1
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 40 | 40
ng/mL | 26.3 [23.9 to 28.9] | 27.2 [25.3 to 29.2]
Statistical Analysis 1: Comparison: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) vs EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca); 39 volunteers qualified for statistical analysis of BE whereas all 40 volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 98.66, 90% CI [93.37 to 104.24] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Mean Area Under the Concentration-time Curve (AUC) of DRSP Incl. Bioequivalence (BE) Evaluation
Description: as for outcome 2
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng∙h/mL
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 40 | 40
ng∙h/mL | 433 [397 to 473] | 447 [417 to 479]
Statistical Analysis 1: Comparison: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) vs EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca); [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 99.45, 90% CI [96.70 to 102.28] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Mean Maximum Concentration (Cmax) of L-5-methyl-THF (Baseline Corrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline corrected Cmax is a measure of the highest measured drug concentration provided solely by the treatment after subtracting endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples, measuring the concentrations of L-5-methyl-THF in each sample and by subtracting the pre-treatment concentration.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Groups:
- L-5-MTHF Ca 0.451 mg (Metafolin): single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca])
Arm/Group | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 41 | 43
nmol/L | 51.7 [47.1 to 56.9] | 48.7 [44.5 to 53.4]
Statistical Analysis 1: Comparison: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); 41 volunteers qualified for statistical analysis of BE whereas all 41 (EE30/DRSP/L-5-MTHF Ca) and 43 (Metafolin) volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 106.19, 90% CI [99.18 to 113.68] — Point estimate for the ratio [(EE30/DRSP/L-5-MTHF Ca) / Metafolin]. Bioequivalence is established if the 90% confidence interval fall within the equivalence interval limits of 80-125%

6. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of L-5-methyl-THF (Baseline Corrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline corrected AUC is a measure of the systemic drug exposure provided by the treatment excluding the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples, measuring the concentrations of L-5-methyl-THF in each sample and by subtracting the pre-treatment concentration.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol∙h/L
Arm/Group | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 41 | 43
nmol∙h/L | 236 [218 to 256] | 239 [221 to 259]
Statistical Analysis 1: Comparison: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 97.98, 90% CI [94.19 to 101.93] — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Mean Maximum Concentration (Cmax) of L-5-methyl-THF (Baseline Uncorrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline uncorrected Cmax is a measure of the highest measured drug concentration including the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples and measuring the concentrations of L-5-methyl-THF in each sample.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 41 | 43
nmol/L | 65.2 [59.3 to 71.6] | 61.8 [56.6 to 67.5]
Statistical Analysis 1: Comparison: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 104.90, 90% CI [98.83 to 111.34] — [estimate comment as in outcome 5, analysis 1]

8. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of L-5-methyl-THF (Baseline Uncorrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline uncorrected AUC is a measure of the systemic drug exposure provided by the treatment including the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples and measuring the concentrations of L-5-methyl-THF in each sample.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol∙h/L
Arm/Group | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 41 | 43
nmol∙h/L | 393 [356 to 435] | 390 [353 to 431]
Statistical Analysis 1: Comparison: EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 99.63, 90% CI [95.73 to 103.69] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of EE
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content
Time Frame: up to 96 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 42 | 42
hour | 2.00 [0.50 to 4.00] | 2.00 [1.00 to 4.00]

10. Secondary Outcome: Mean Area Under the Concentration-time Curve From Administration up to 72h AUC(0-72h) of DRSP
Description: as for outcome 2
Time Frame: up to 72 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng∙h/mL
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 40 | 40
ng∙h/mL | 352 [323 to 383] | 366 [346 to 388]
Statistical Analysis 1: Comparison: EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) vs EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca); 38 volunteers qualified for statistical analysis of BE whereas all 40 volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 99.57, 90% CI [97.32 to 101.87] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of DRSP
Description: as for outcome 9
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 40 | 40
hour | 1.50 [1.00 to 3.00] | 1.50 [0.50 to 3.00]

12. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of L-5-methyl-THF
Description: as for outcome 9
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 41 | 43
hour | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.50]

ADVERSE EVENTS:
Groups:
- L-5-MTHF Ca 0.451mg (Metafolin): single oral administration of 1 coated tablet SHT04532C, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca])
Arm/Group | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451mg (Metafolin)
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 27/44 | 31/43 | 16/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EE 0.03 mg/DRSP 3 mg (Yasmin, BAY86-5131) (N=44) | EE 0.03mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE30/DRSP/L-5-MTHF Ca) (N=43) | L-5-MTHF Ca 0.451mg (Metafolin) (N=43)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 9 (9) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 9 (9) | 12 (12) | 7 (7)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 4 (4) | 6 (7)
Syncope vasovagal (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 3 (3) | 7 (8) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI (principal investigator) of CRO (contract research organization) will refrain from publishing any data or information generated or derived as a result of the performance of the Services.